CLINICAL TRIAL: NCT00950430
Title: Brain Amyloid Imaging With Pittsburgh Compound B in Normal Aging, Mild Cognitive Impairment, and Dementia
Brief Title: Imaging of Brain Amyloid Plaques in the Aging Population
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Val Lowe, Consultant - Diagnostic Radiology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-005553; U01AG006786 (NIH); R01AG011378 (NIH)
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer's Disease; Dementia With Lewy Bodies; Frontotemporal Dementia; Vascular Dementia
Keywords: Imaging; PET; PiB; FDG; MCI; Dementia; Alzheimer's Disease; Brain Amyloid
MeSH Terms: conditions — Alzheimer Disease; Lewy Body Disease; Frontotemporal Dementia; Dementia, Vascular; Dementia | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole; tau Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PiB PET, FDG PET, Tau PET (Experimental)
  Interventions: Drug: Pittsburgh Compound B (C-11 PiB); Drug: F-18 FDG; Drug: Tau (18-F-AV-1451)

INTERVENTIONS:
Drug: Pittsburgh Compound B (C-11 PiB) — Repeat these scans approximately every 24-30 months for up to 10 years in those with all three PETs or 20 years in those with only PiB PET and FDG PET. A second PiB PET, TAU PET and/or FDG PET may be administered within a year if needed to ensure a completed exam for analysis in the rare case of exam failure or data loss.
Drug: F-18 FDG — Repeat these scans approximately every 24-30 months for up to 10 years in those with all three PETs or 20 years in those with only PiB PET and FDG PET. A second PiB PET, TAU PET and/or FDG PET may be administered within a year if needed to ensure a completed exam for analysis in the rare case of exam failure or data loss.
Drug: Tau (18-F-AV-1451) — 1. PIB PET scan, Tau PET scan and/or FDG PET scan
  2. Repeat these scans approximately every 24-30 months for up to 10 years in those with all three PETs or 20 years in those with only PiB PET and FDG PET. A second PiB PET, TAU PET and/or FDG PET may be administered within a year if needed to ensure a completed exam for analysis in the rare case of exam failure or data loss. ECG will be performed on subjects who have not had previous ECG test at Mayo to rule out prolonged QT interval prior to PET TAU scan.

SUMMARY:
This is a prospective, open label, non-therapeutic, diagnostic imaging study. The purpose of this study is to utilize Pittsburgh Compound B positron emission imaging (PiB PET) to ascertain the relationship between change in amyloid burden over time, and concurrent change in clinical status.

DETAILED DESCRIPTION:
Identification of risk factors and biomarkers of neurodegenerative disease is essential in caring for the growing numbers of elderly. Imaging biomarkers provide non-invasive ways to look at brain function. A new PET imaging agent, Pittsburgh Compound B (PiB), that identifies brain amyloid is an exciting development in brain imaging that needs to be studied. We plan to study this imaging technique in normal volunteers and patients with a variety of neurodegenerative diseases to determine its utility. Long term followup of these subjects will allow us to understand the predictive ability of this new test.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-100
* Subjects who have completed or are scheduled to undergo the neurological evaluation procedures in the Mayo Clinic Study of Aging, Mayo ADRC, or Mayo neurodegenerative disease clinics.

Exclusion Criteria:

* Subjects unable to lie down without moving for 10 minutes
* Women who are pregnant or cannot stop breast feeding for 24 hours at the time of scanning
* Claustrophobic patients unable to tolerate the scans
* Standard safety exclusionary criteria for MRI such as metallic foreign bodies, pacemaker, etc.

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2008-04; Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
To understand the predictive ability of PiB PET imaging for neurodegenerative diseases. | up to 20 years

SECONDARY OUTCOMES:
Using PiB-PET, to ascertain cross-sectionally the magnitude and the spatial distribution of amyloid deposition in the brain in subjects who are clinically classified as CN, MCI, and demented. | up to 20 years
To identify the relationship between amyloid burden and the risk of progression from CN at baseline to MCI. | up to 20 years
To identify the relationship between amyloid burden and the risk of progression from MCI at baseline to dementia. | up to 20 years
To measure longitudinal change in amyloid burden and cognition and characterize the correlation between change on serial PiB-PET measures vs. FDG measures and concurrent change on continuous measures of cognitive performance. | up to 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Val Lowe, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No